CLINICAL TRIAL: NCT02581891
Title: Managing Neovascular Age-related Macular Degeneration (nAMD) Over 2 Years With a Treat and Extend (T&E) Regimen of 2 mg Intravitreal Aflibercept - a Randomized, Open-label, Active-controlled, Parallel-group Phase IV/IIIb Study (ARIES)
Brief Title: Managing Neovascular (Known as "Wet") Age-related Macular Degeneration Over 2 Years Using Different Treatment Schedules of 2 mg Intravitreal Aflibercept Injected in the Eye
Acronym: ARIES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17508; 2014-003132-39 (EudraCT Number)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Macular Degeneration
Keywords: Neovascular age-related macular degeneration; nAMD)
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Early-start T&E / Arm 1 (Experimental): Early-start T&E arm: test group, early treatment individualization
  Interventions: Drug: Eylea (Intravitreal Aflibercept, VEGF Trap-Eye, BAY86-5321)
- Late-start T&E / Arm 2 (Active Comparator): Late-start T&E arm; per label, control group, treatment individualization after Year 1
  Interventions: Drug: Eylea (Intravitreal Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Intravitreal Aflibercept, VEGF Trap-Eye, BAY86-5321) — 3 monthly doses followed by individualized treatment intervals of between 8 to16 weeks based on protocol-defined anatomical criteria
  Arms: Early-start T&E / Arm 1
Drug: Eylea (Intravitreal Aflibercept, VEGF Trap-Eye, BAY86-5321) — 3 monthly doses followed by five 8-weekly doses (5 x 2Q8), then by individualized treatment intervals of between 8 to 16 weeks based on protocol-defined anatomical criteria
  Arms: Late-start T&E / Arm 2

SUMMARY:
This study aims to evaluate the optimal use, efficacy, and safety of a Treat-and-Extend regimen with aflibercept in subjects with nAMD.

DETAILED DESCRIPTION:
The T&E dosing regimen for nAMD has emerged as a preferred regimen for many treating physicians aiming at maximizing outcomes by proactively treating the subject at each visit and by extending the treatment interval (if extension criteria are met), thus limiting visits, monitoring, and injections.

To this day, there is limited evidence available addressing the question of what are useful intervals for treating and monitoring, how do they differ among subjects, and how are retreatment criteria applied to achieve long-term desirable outcomes in real-life practice. This study is designed to evaluate the optimal use, efficacy, and safety of the T&E regimen with intravitreal aflibercept in subjects with nAMD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 50 years of age.
* Active primary subfoveal CNV lesions secondary to nAMD, including juxtafoveal lesions that affect the fovea as evidenced by FA in the study eye. Patients with polypoidal choroidal vasculopathy or retinal angiomatous proliferation are eligible to participate in the study, and their condition should be captured in the eCRF.
* ETDRS BCVA of 73 to 25 letters (20/40 to 20/320 Snellen equivalent) in the study eye.
* The area of CNV must occupy at least 50% of the total lesion.

Exclusion Criteria:

* Any prior ocular (in the study eye) or systemic treatment or surgery for nAMD, except dietary supplements or vitamins.
* Any prior or concomitant therapy with another investigational agent to treat nAMD in the study eye.
* Prior treatment with anti-VEGF agents as follows:
* Prior treatment with anti-VEGF therapy in the study eye is not allowed
* Prior treatment with anti-VEGF therapy in the fellow eye with an investigational agent (not approved, e.g. bevacizumab) within the last 3 months before the first dose in the study. Such treatment will also not be allowed during the study. Prior treatment with an approved anti-VEGF therapy in the fellow eye is allowed.
* Prior systemic anti-VEGF therapy, investigational or approved, within the last 3 months before the first dose in the study, and such treatment will not be allowed during the study.
* Total lesion size >12 disc areas (30.5 mm2, including blood, scars and neovascularization) as assessed by FA in the study eye.
* Subretinal hemorrhages that are either 50% or more of the total lesion area, or if the blood is under the fovea and is 1 or more disc areas in size in the study eye. (If the blood is under the fovea, then the fovea must be surrounded by 270 degrees by visible CNV).
* Scar or fibrosis making up >50% of the total lesion in the study eye.
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Presence of retinal pigment epithelial tears or rips involving the macula in the study eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Australia (5):
  - Strathfield, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
  - Launceston
- Canada (3):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Boisbriand, Quebec
- France (2):
  - Créteil
  - Nice
- Germany (8):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Hanover, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Sulzbach, Saarland
  - Chemnitz, Saxony
  - Berlin
- Hungary (4):
  - Budapest
  - Debrecen
  - Pécs
  - Szombathely
- Italy (3):
  - Rome, Lazio
  - Milan, Lombardy
  - Padua, Veneto
- Spain (3):
  - Oviedo, Principality of Asturias
  - Madrid
  - Zaragoza
- United Kingdom (5):
  - Canterbury, Kent
  - Bristol
  - Liverpool
  - London
  - Oxford

REFERENCES:
- [Result] Wolf S, Holz FG, Midena E, Souied EH, Lambrou G, Machewitz T, Allmeier H, Mitchell P; ARIES Study Investigators. Patients with Neovascular Age-Related Macular Degeneration Requiring Intensive Intravitreal Aflibercept Treatment: An ARIES Post Hoc Analysis. Ophthalmol Ther. 2022 Oct;11(5):1793-1803. doi: 10.1007/s40123-022-00541-8. Epub 2022 Jul 12. PMID 35821380
- [Result] Chaudhary V, Holz FG, Wolf S, Midena E, Souied EH, Allmeier H, Lambrou G, Machewitz T, Mitchell P; ARIES study investigators. Association Between Visual Acuity and Fluid Compartments with Treat-and-Extend Intravitreal Aflibercept in Neovascular Age-Related Macular Degeneration: An ARIES Post Hoc Analysis. Ophthalmol Ther. 2022 Jun;11(3):1119-1130. doi: 10.1007/s40123-022-00491-1. Epub 2022 Mar 18. PMID 35303285
- [Result] Tuerksever C, Somfai GM, Oesch S, Machewitz T, Hasler PW, Zweifel S. Hypothetical Switch of Anti-Vascular Endothelial Growth Factor in Neovascular Age-Related Macular Degeneration: An ARIES Post Hoc Analysis. Ophthalmol Ther. 2022 Apr;11(2):613-627. doi: 10.1007/s40123-021-00448-w. Epub 2022 Jan 23. PMID 35066801
- [Derived] Krieger N, Chen JT, Testa C, Diez Roux A, Tilling K, Watkins S, Simpkin AJ, Suderman M, Davey Smith G, De Vivo I, Waterman PD, Relton C. Use of Correct and Incorrect Methods of Accounting for Age in Studies of Epigenetic Accelerated Aging: Implications and Recommendations for Best Practices. Am J Epidemiol. 2023 May 5;192(5):800-811. doi: 10.1093/aje/kwad025. PMID 36721372
- [Derived] Mitchell P, Holz FG, Hykin P, Midena E, Souied E, Allmeier H, Lambrou G, Schmelter T, Wolf S; ARIES study investigators. EFFICACY AND SAFETY OF INTRAVITREAL AFLIBERCEPT USING A TREAT-AND-EXTEND REGIMEN FOR NEOVASCULAR AGE-RELATED MACULAR DEGENERATION: The ARIES Study: A Randomized Clinical Trial. Retina. 2021 Sep 1;41(9):1911-1920. doi: 10.1097/IAE.0000000000003128. PMID 33782365
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/17508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 19-Nov-2015 (First Patient First Visit) to 26-Apr-2019 (Last Patient Last Visit).
Pre-assignment Details: A total of 443 participants were screened in this study. Of these, 156 participants were screening failures and did not enter the treatment period. Of the 287 treated participants, 16 were treated during the initiation phase, but were not randomized to a treatment arm after the initiation phase.
Groups:
- Early-start T&E Arm: All participants during the initiation phase received Aflibercept (Eylea, BAY86-5321) 3 doses at Weeks 0, 4, and 8 followed by one dose 2Q8 (2 mg administered every 8 weeks) at Week 16. From Week 16 to Week 104 participants randomized to Early-start T&E arm (Treat and Extend arm) received treatment in individualized intervals of between 8 to16 weeks based on anatomical criteria.
- Late-start T&E Arm: All participants during the initiation phase received Aflibercept (Eylea, BAY86-5321) 3 doses at Weeks 0, 4, and 8 followed by one dose 2Q8 (2 mg administered every 8 weeks) at Week 16. From Week 16 participants randomized to Late-start T&E arm received four 2Q8 injections. In Year 2 starting at Week 48, participants received treatment in individualized intervals of between 8 to16 weeks based on anatomical criteria.
Period: Overall Study
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Started (Randomized) | 135 | 136
Completed Treatment | 120 | 117
Completed (Completed Study) | 119 | 117
Not Completed | 16 | 19
Not completed — Adverse Event | 4 | 6
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Other Reasons | 3 | 1
Not completed — Discontinued during followup | 1 | 0

BASELINE CHARACTERISTICS:
Population: All 271 participants were included in the SAF (287), who received any study drug in this study.
  269 participants were included in the FAS, excluding 16 participants who were treated but not randomized and 1 participant in each treatment arm from SAF.
  Of the 269 participants in FAS, 59 participants in total were excluded from the PPS (210).
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-start T&E Arm | Late-start T&E Arm | Total
Number analyzed (Participants) | 135 | 136 | 271
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76 (8.8) | 76.9 (8.2) | 76.5 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 73 | 154
  Male | 54 | 63 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 126 | 122 | 248
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 131 | 127 | 258
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 8 | 9
Baseline BCVA letters scores (study eye) [Mean (Standard Deviation); unit: letters] — BCVA = best corrected visual acuity Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
  letters
    number analyzed (Participants) | 106 | 104 | 210
    (all) | 60.2 (12.1) | 61.3 (10.8) | 60.8 (11.4)
Baseline CRT [Mean (Standard Deviation); unit: μm] — CRT = central retinal thickness Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
  μm
    number analyzed (Participants) | 106 | 104 | 210
    (all) | 443.7 (120.0) | 448.3 (133.1) | 446.0 (126.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in BCVA as Measured by the ETDRS Letter Score
Description: BCVA (best corrected visual acuity) was measured by the ETDRS (Early Treatment Diabetic Retinopathy Study) letter score of 73 to 25 (= Acuity of 20/40 to 20/320) in the study eye at 4 meters; a higher score represents better functioning.
Time Frame: From Week 16 to Week 104
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Letters correctly read | -2.1 (11.4) | -0.4 (8.4)
Statistical Analysis 1: Comparison: Early-start T&E Arm vs Late-start T&E Arm; Test type: Non-Inferiority — The non-inferiority margin is set to 5 letters; p = 0.0162, ANCOVA; LS mean difference = -2.0199, 95% CI 2-sided [-4.7470 to 0.7073], Standard Error of Mean 1.3833

2. Secondary Outcome: Percentage of Participants Maintaining Vision (<3 Lines Loss) at Week 104 Compared With Baseline
Description: Participants maintained 3 lines (15 letters) vision loss in BCVA (Best-corrected visual acuity) as measured by the ETDRS (Early Treatment Diabetic Retinopathy Study) letter.
Time Frame: at Week 104
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Number; unit: Percentage
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Percentage | 93.4 | 96.2

3. Secondary Outcome: Change in BCVA From Baseline to Week 52, Baseline to Week 104, and Week 16 to Week 52
Description: as for outcome 1
Time Frame: from baseline to Week 52, baseline to Week 104, and Week 16 to Week 52
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Letters
  From baseline to Week 52 | 7.8 (9.4) | 10.2 (9.3)
  From baseline to Week 104 | 4.3 (13.4) | 7.9 (11.9)
  Week 16 | 66.7 (13.0) | 69.6 (11.6)
  From Week 16 to Week 52 | 1.3 (6.4) | 2.0 (5.3)

4. Secondary Outcome: Percentage of Participants Maintaining Vision (<3 Lines Loss) at Week 52 Compared With Baseline
Description: as for outcome 2
Time Frame: At week 52
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Number; unit: Percentage
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Percentage | 100.0 | 100.0

5. Secondary Outcome: Percentage of Participants Gained 3-line at Week 52 and Week 104 Compared With Baseline
Description: Participants gained 3 lines (15 letters) in BCVA (Best-corrected visual acuity) as measured by the ETDRS (Early Treatment Diabetic Retinopathy Study) letter.
Time Frame: At Week 52 and Week 104
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Number; unit: Percentage
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Percentage
  Week 52 | 19.8 | 27.9
  Week 104 | 18.9 | 22.1

6. Secondary Outcome: Change in Central Retinal Thickness (CRT)
Description: CRT were evaluated using spectral domain Optical coherence tomograph (OCT).
Time Frame: From baseline to Week 52, baseline to Week 104, Week 16 to Week 52, and Week 16 to Week 104
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
μm
  From baseline to Week 52 | -164.9 (117.3) | -167.1 (117.1)
  From baseline to Week 104 | -161.6 (135.6) | -158.6 (125.1)
  Week 16 | 321.4 (93.4) | 322.5 (104.0)
  From Week 16 to Week 52 | -28.5 (56.3) | -28.7 (54.0)
  From Week 16 to Week 104 | -25.1 (68.9) | -20.2 (70.0)

7. Secondary Outcome: Number of Study Drug Injections From Baseline to Week 52 and Baseline to Week 104
Time Frame: At Week 52 and Week 104
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
injections
  Week 52 | 7.1 (0.8) | 8.0 (0.2)
  Week 104 | 12.0 (2.3) | 13.0 (1.8)

8. Secondary Outcome: Duration of Last Treatment Interval
Time Frame: Early-Start T&E: from week 16 up to Week 104 or early termination; Late-Start T&E: From end of Year 1 up to Week 104 or early termination
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
Weeks | 11.5 (3.7) | 11.4 (3.7)

9. Secondary Outcome: Percentage of Participants Requiring Retreatment at 8 Weeks, 10 Weeks, 12 Weeks, 14 Weeks, and 16 Weeks as the Last Treatment Interval
Time Frame: at 8 weeks, 10 weeks, 12 weeks, 14 weeks, and 16 weeks
Population: PPS (Per-protocol set): all participants in the FAS (full analysis set) without any major protocol deviation.
Measure: Number; unit: percentage
Arm/Group | Early-start T&E Arm | Late-start T&E Arm
Number analyzed (Participants) | 106 | 104
percentage
  <8 weeks | 5.7 | 7.7
  8 weeks | 27.4 | 29.8
  10 weeks | 19.8 | 10.6
  12 weeks | 8.5 | 13.5
  14 weeks | 8.5 | 11.5
  16 weeks | 25.5 | 25.0
  >16 weeks | 4.7 | 1.9

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were AEs that started after the first application of aflibercept up to 30 days after last study drug Injection in the study. TEAEs were collected from Week 0 till End of study/Week 104 or early termination.
Description: Below adverse events were reported based on Safety Analysis Set (SAF), which included all participants who received any study drug in this study. The participants who dropped out after start of treatment before randomization were not allocated to a treatment arm, but were included in this SAF.
Groups:
- Treated, But Not Randomized: Participants were treated during the initiation phase, received Aflibercept (Eylea, BAY86-5321) 3 doses at Weeks 0, 4 and 8 followed by one dose 2Q8 (2 mg administered every 8 weeks)at Week 16, but were not randomized to a treatment arm after the initiation phase.
Arm/Group | Early-start T&E Arm | Late-start T&E Arm | Treated, But Not Randomized
All-Cause Mortality (participants affected / at risk) | 3/135 | 4/136 | 0/16
Serious Adverse Events (participants affected / at risk) | 29/135 | 35/136 | 3/16
Other Adverse Events (participants affected / at risk) | 93/135 | 80/136 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-start T&E Arm (N=135) | Late-start T&E Arm (N=136) | Treated, But Not Randomized (N=16)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal artery embolism (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 5 (5) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-start T&E Arm (N=135) | Late-start T&E Arm (N=136) | Treated, But Not Randomized (N=16)
Blepharitis (Eye disorders) | 2 (6) | 11 (25) | 0 (0)
Cataract (Eye disorders) | 9 (14) | 8 (13) | 0 (0)
Cataract nuclear (Eye disorders) | 2 (4) | 7 (16) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 20 (26) | 18 (20) | 0 (0)
Corneal erosion (Eye disorders) | 5 (6) | 2 (3) | 1 (1)
Dry eye (Eye disorders) | 6 (11) | 11 (18) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Macular degeneration (Eye disorders) | 6 (6) | 5 (5) | 1 (1)
Punctate keratitis (Eye disorders) | 10 (23) | 5 (9) | 1 (1)
Retinal haemorrhage (Eye disorders) | 4 (4) | 6 (7) | 2 (2)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Visual acuity reduced (Eye disorders) | 21 (24) | 17 (19) | 1 (1)
Visual impairment (Eye disorders) | 8 (11) | 4 (4) | 0 (0)
Vitreous floaters (Eye disorders) | 8 (8) | 4 (5) | 0 (0)
Vitreous adhesions (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 7 (7) | 5 (5) | 0 (0)
Retinal pigment epithelial tear (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 15 (15) | 14 (14) | 1 (1)
Macular fibrosis (Eye disorders) | 2 (2) | 6 (6) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 11 (12) | 12 (13) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (21) | 17 (22) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 13 (15) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT02581891/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT02581891/SAP_001.pdf